CLINICAL TRIAL: NCT04264923
Title: Pilot Study: Quality Evaluation of Stool Samples Collected for Microbiome Analysis Using the HyGIeaCare Prep
Brief Title: Evaluation of Stool Microbiome Using HyGIeaCare Prep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HyGIeaCare, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HGP-0002
Record Dates: First submitted 2019-07-24; First posted 2020-02-11 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2019-06

CONDITIONS: Stool Microbiome

STUDY DESIGN:
Intervention Model Description: Patients between 18 and 80 years old who do not have any known health issues and who have not taken antibiotics within the last two months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All patients enrolled (Experimental): All patients enrolled with receive the HyGIeaCare Prep with a new lab sampling technique to be used on all patients enrolled in the study.
  Interventions: Other: HyGIeaCare Prep

INTERVENTIONS:
Other: HyGIeaCare Prep — Each patient will have up to 5 stool specimens for evaluation by a lab for microbial contents.
  Other Names: Stool sample evaluation

SUMMARY:
Stool samples will be collected before and during the HyGIeaCare procedure and the samples will be sent for microbiome evaluation.

DETAILED DESCRIPTION:
Patients will have the HyGIeaCare procedure as originally prescribed by their physician. Before and during the procedure stool samples will be collected and sent to a lab for microbiome evaluation.

It is anticipated that stool samples collected from the HyGIeaCare prep will provide more microbiological and biochemical information on the gut interior than using traditional stool samples.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's age is between 18 and 80 years old scheduled for elective screening or polyp surveillance indicated colonoscopy
2. Patient does not have any known health issues (as listed in exclusion criteria)
3. Patient had not taken antibiotics within the last 2 months

Exclusion Criteria:

1. Patient has functional bowel disorders characterized by alternating bowel habits (diarrhea/constipation), chronic diarrhea or chronic constipation (requiring pharmacologic prescription treatment)
2. Patient has secondary constipation (colonic obstruction, medications, metabolic cause)
3. Patient has any other condition that, in the opinion of the investigator, may adversely affect the compliance or safety of the patient or would limit the patient's ability to complete the study
4. Patient has any of the contraindications listed below:

   1. Cardiac: Congestive heart failure (NYHA class III or IV or EF <50%)
   2. GI: Intestinal perforation, carcinoma of the rectum, fissures or fistula, severe hemorrhoids, abdominal hernia, recent colon or rectal surgery, or abdominal surgery, inflammatory bowel disease. History of gastrointestinal surgery- (small bowel, colon. Bariatric surgery)
   3. GU: Renal insufficiency (CC < 60 ml/min/173m2), cirrhosis with ascites
   4. Abdominal surgery within the last 6 months
   5. Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Microbial classification | 6 months
  The number of genes present will be counted
Diversity between stool and colon effluent samples | 6 months
  Alpha diversity by Shannon diversity index, presence and number of taxa to be documented
Inner diversity of samples | 6 months
  ANOVA test will be used to acknowledge differences between samples, presence and number of taxa to be documented
Contribution of the variables to samples' diversity | 6 months
  Principal component analysis (PCoA) will be used to mark significant differences between the samples, taxa will be identified by presence, percentage of sample will be documented

SECONDARY OUTCOMES:
Functional genes analysis | 6 months
  The presence of genes known to represent biochemical functions will be counted and documented
Biosynthetic gene clusters | 6 months
  Groups of genes with known biosynthetic functions and found to be clustered will be counted and documented together in the different samples

CONTACTS AND LOCATIONS:
Overall Officials: David A Johnson, MD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- HyGIeaCare Center, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Initially the data will be used internally.